CLINICAL TRIAL: NCT06274762
Title: Breast Cancer Awareness of Women With Visual Impairment and Self-administered Health Belief Model-Based Education Effect on Breast Examination Skills
Brief Title: Visually Impaired Women Model-based Cancer Education and Breast Self-examination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Seval Saray Demir, PhD student, Marmara University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MARU-SBF-ROKÇ-01
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Awareness and BSE in Visually Impaired Women
Keywords: Visually impaired women; breast self-examination; breast cancer
MeSH Terms: conditions — Breast Self-Examination; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: There is an experimental group of 45 visually impaired women aged 20-69 and a control group of 45. Randomization was not possible. Blinding could not be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A pre-test will be conducted to determine socio-demographic data and to assess breast cancer awareness (champion health belief model scale). Experimental and control groups will be formed. The 45 people in the experimental group will be divided into 5 groups of 8 people. Each group will receive 45 minutes of theoretical training and 60 minutes of BSE application and will be explained and applications will be provided on the model. Question - Answer - 20 minutes will be allocated for feedback. 5 groups will be allocated one day each.4 weeks after the training, the experimental group will be called again in 5 groups and the champion health belief model scale will be repeated, they will be asked to perform the BSE application on the model and evaluation will be made according to the BSE evaluation form prepared by the researcher. 6 months after the study, the whatsapp group will be questioned about whether individuals have BSE.
  Interventions: Other: Training and BSE application on a model
- Control Group (Active Comparator): A pre-test will be conducted to determine socio-demographic data and to assess breast cancer awareness (champion health belief model scale). Experimental and control groups will be formed.The control group will not be intervened until the study is over.
  Interventions: Other: Training and BSE application on a model

INTERVENTIONS:
Other: Training and BSE application on a model — A breast cancer awareness training designed according to the headings of sensitivity, seriousness, benefit, obstacle perception, health motivation and self-efficacy, which are the steps of the health belief model, followed by applied BSE on a model.
  Other Names: Health Belief Model Based Education

SUMMARY:
The aim of our study was to raise awareness among visually impaired women, who are in the vulnerable group, about breast cancer, which ranks first among female cancers, and to teach breast self-examination.

DETAILED DESCRIPTION:
Cancer ranks second after cardiovascular diseases among the causes of death in the world and in our country and it is predicted that by 2030 this situation will change due to changing living and environmental conditions and cancer will take the first place. Breast cancer is the most common type of cancer among female cancers. Breast cancer is a type of cancer that can be prevented and treated if diagnosed early. For this reason, screening programs have been developed to prevent breast cancer and these screening programs include breast self-examination (BSE), clinical breast examination and mammography. These screening programs, which are also accepted in our country, include all women between the ages of 20-69. should be included. However, 11% of breast cancer cases are diagnosed at a distant stage. Disability for women, it affects their access to health services; people's perceptions of disability, inappropriate health services facilities and equipment, stereotypes and discrimination, economic inadequacy, negative treatment from staff, unequal allocation of time and money within the household for their care, limited health service coverage and lack of disability-related education, sensitization or recognition of women as a person in need of sexual and reproductive health care impede women's seeking, use and access to health care. However, every woman has the right to regular gynecological examinations and good care. In our study, the breast cancer awareness of visually impaired women and the effect of training based on the health belief model on their ability to perform breast self-examination will be evaluated. The population of the study consists of visually impaired women between the ages of 20-69. The sample of the study was calculated based on Cohen's effect size study.

Taking d (effect size) as 0.8, α= 0.05 and power as 0.95, the experimental group was determined as 42 and the control group as 42 people. G power 3.1 program was used in the calculations. Considering the problems that may occur during the research process, 45 in the experimental group and 45 in the control group, a total of 90 people constitute the sample of the study. As data collection tools; a questionnaire form including sociodemographic data created by the researchers, Champion's Health Belief Model Scale and KKMM Skill Checklist on Model will be used. The data will be analyzed with descriptive analyses in SPSS program and pre-test - post-test comparative analyses will be performed to determine the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being visually impaired
* Volunteering to participate in research
* Not having any disability other than visual impairment
* Being knowledgeable individuals who can communicate
* Not being diagnosed with breast cancer

Exclusion Criteria:

* Not being willing to participate in the research
* Not filling out research-related forms completely
* Abandoning the study at any time during the research

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Visually impaired women aged 20-69
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Champion health belief model scale | two weeks
  The scale evaluates the individual's judgment about breast cancer and general health, including "sensitivity", "importance/seriousness" and "health motivation", "obstacles", "benefits" regarding BSE, "self-efficacy/confidence", "benefits" regarding mammography. " and "obstacles" dimensions. Which dimensions of the scale will be used varies depending on the purpose of the study and the characteristics of the study group. A 5-point Likert type scaling method ranging from 1 to 5 was used to evaluate the scale. Each dimension of the scale is evaluated separately and is not combined into a single total score. Accordingly, points equal to the number of dimensions used are obtained for each individual. Although completing the scale depends on which dimensions are used, it takes approximately 12-15 minutes when all of them are used. The scale consists of 36 items and 6 factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No